CLINICAL TRIAL: NCT01396681
Title: Phase Ⅱ Trial of Postoperative Adjuvant Gemcitabine and Cisplatin Chemotherapy Followed by Chemoradiation With Gemcitabine in Patients With Resected Pancreatic Cancer
Brief Title: Adjuvant Gemcitabine and Cisplatin Followed by Chemoradiation for Resected Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Seock-Ah Im, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-0412-138-006
Record Dates: First submitted 2011-07-01; First posted 2011-07-19 (Estimated); Last update posted 2011-07-19 (Estimated); Status verified 2011-07

CONDITIONS: Pancreatic Cancer
Keywords: resected pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: gemcitabine and cisplatin — The study consists of three phases; Induction chemotherapy phase:Starting 4~8 weeks after R0 resection of pancreatic cancer. Gemcitabine: 1200mg/㎡ (Day 1, 8), cisplatin 60mg/㎡ (Day 1) every 3 weeks for 2 cycles. Chemoradiotherapy phase: Starting 1-2 weeks after completion of induction chemotherapy (within 5 weeks after D1 of 2nd cycle of induction chemotherapy), no later than 16 weeks after operation. Gemcitabine 300mg/㎡ weekly for 5 weeks throughout RT period. Radiotherapy: 50.4Gy at 1.8Gy/Fx, for 28 Fx (Field reduction at 45Gy) for 5.5 pweeks. Maintenance chemotherapy phase: Within 4 weeks after completion of chemoradiotheray, no later than 6 weeks after completion of chemoradiotherapy Gemcitabine: 1200mg/㎡ (Day 1, 8) every 3 weeks, for 4 cycles

SUMMARY:
This is a phase Ⅱ Trial of Postoperative Adjuvant Gemcitabine and Cisplatin Chemotherapy Followed by Chemoradiation With Gemcitabine in Patients With Resected Pancreatic Cancer.

DETAILED DESCRIPTION:
The primary study objective is to evaluate recurrence/metastasis free survival at 12 months with postoperative adjuvant treatment incorporating gemcitabine plus cisplatin chemotherapy followed by chemoradiation with gemcitabine followed by maintenance chemotherapy with gemcitabine.

ELIGIBILITY:
Inclusion Criteria:

1. Give written informed consent prior to study specific screening procedures, with the understanding that the patient has the right to withdraw from the study at any time, without prejudice.
2. Be between 18 and 75 years of age.
3. Patients who are ambulatory and have a ECOG Performance Status of 0-2.
4. Histologically confirmed pancreatic adenocarcinoma.
5. Received curative resection (R0 resection) of stage 1b ~ 2b pancreatic cancer (according to AJCC staging, 6th edition - Appendix 1), no more than 8 weeks has elapsed since the time of operation.
6. WBC at least 3,000/mm3 OR Absolute neutrophil count at least 1,500/mm3. Platelet count at least 100,000/mm3.
7. Bilirubin less than 2.0 mg/dL, AST less than 3 times upper limit of normal (ULN).

Serum creatinine no greater than 1.5 times ULN.

Exclusion Criteria:

1. Pregnant or lactating woman.
2. Woman of childbearing potential with either a positive or no pregnancy test at baseline.
3. Woman of childbearing potential not using a reliable and appropriate contraceptive method (postmenopausal women must have been amenorrheic for at least 12 months to be considered of non-childbearing potential).
4. Sexually active males unwilling to practice contraception during the study.
5. Prior chemotherapy for the treatment of pancreatic carcinoma.
6. Radiotherapy incorporating radiation fields of more than 25% of active bone marrow.
7. History of another malignancy within the last five years except cured basal cell carcinoma of skin and cured carcinoma in-situ of uterine cervix.
8. Clinically significant cardiac disease (e.g. congestive heart failure, symptomatic coronary artery disease, and cardiac arrhythmias not well controlled with medication).
9. Participation in any investigational drug study within four weeks preceding the start of study treatment.
10. Serious, uncontrolled, intercurrent infection(s).
11. Other significant medical conditions that would, in the judgment of the investigator, make administration of study drug unsafe.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2004-12; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
recurrence/metastasis free survival | 24 months

SECONDARY OUTCOMES:
2 year survival rate | 24 months
Overall survival | 24 months
recurrence free survival | 24 months
  Median recurrence free survival time
Safety and tolerability | 24 months
  patients who experienced grade 3-4 toxicity by RECIST criteria

CONTACTS AND LOCATIONS:
Overall Officials: Seock-Ah Im, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (2):
- South Korea (2):
  - Seoul National University Bundang Hospital, Seongnam
  - Seoul National University Hospital, Seoul